CLINICAL TRIAL: NCT03056989
Title: A Phase 1, Single-Center, Open-Label Safety Study of SPX-101 Inhalation Solution in Subjects With Cystic Fibrosis
Brief Title: A Safety Study of SPX-101 Inhalation Solution in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spyryx Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPX-101-CF-102
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPX-101 Low Dose (Experimental): Inhalation Solution twice daily for 7 days.
  Interventions: Drug: SPX-101
- SPX-101 Mid Dose (Experimental): Inhalation Solution twice daily for 7 days.
  Interventions: Drug: SPX-101
- SPX-101 High Dose (Experimental): Inhalation Solution twice daily for 7 days.
  Interventions: Drug: SPX-101

INTERVENTIONS:
Drug: SPX-101 — Inhalation solution twice daily for 7 days.

SUMMARY:
Ascending dose, 7-day, open label safety trial of SPX-101 Inhalation Solution in adult subjects with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* FEV1 ≥ 40% predicted normal
* Stable CF lung disease
* Non-pregnant, non-lactating females

Exclusion Criteria:

* Significant unstable co-morbidities within 28 days of screening as judged by the Investigator.
* Has received an investigational drug within the past 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Day 1 through Day 15

SECONDARY OUTCOMES:
Relative change from baseline through Day 8 in percent predicted FEV1 | Screening and Day 1 through Day 8
Change from baseline through Day 8 in clinical laboratory tests | Screening and Day 1 through Day 8
  Chemistry, Hematology, Urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Tullis, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- Saint Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Couroux P, Farias P, Rizvi L, Griffin K, Hudson C, Crowder T, Tarran R, Tullis E. First clinical trials of novel ENaC targeting therapy, SPX-101, in healthy volunteers and adults with cystic fibrosis. Pulm Pharmacol Ther. 2019 Oct;58:101819. doi: 10.1016/j.pupt.2019.101819. Epub 2019 Jul 11. PMID 31302339